CLINICAL TRIAL: NCT04648228
Title: Integrated Treatment for Veterans With Co-Occurring Chronic Pain and Opioid Use Disorder
Brief Title: Pain and Opioids: Integrated Treatment In Veterans
Acronym: POSITIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Utah (Other); Johns Hopkins University (Other); Duke University (Other); Vanderbilt University (Other); Biomedical Research Institute of New Mexico (Other); Seattle Institute for Biomedical and Clinical Research (Other); Queen's University, Belfast (Other); University of California, San Francisco (Other); San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1507090; 1UG3DA051241-01 (NIH); A20-0217 (Other: Cayuse Project Number)
Record Dates: First submitted 2020-06-18; First posted 2020-12-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Opioid-use Disorder; Opioids; Harmful Use
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This trial will determine the efficacy of an integrated Acceptance and Commitment Therapy and Mindfulness-Based Relapse Prevention (ACT+MBRP) treatment program for veterans with co-occurring chronic pain and opioid use disorder (OUD) who are prescribed buprenorphine, compared to an education control (EC) consisting of pain, opioid, and buprenorphine education. To test the efficacy of ACT + MBRP compared to EC with regard to primary and secondary outcomes, participants will be randomized to one of 2 treatment arms and followed for a total of 15 months (3-month active treatment period, 6 month follow-up, 12 month follow-up). All study treatments will be delivered via the VA Video Connect telehealth platform.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigators will be blinded. Co-investigators and study physicians involved in the treatment and control conditions will not be blinded, as these individuals will handle the delivery of treatment. The study coordinators located within each VA will not be blinded, as they will be involved in coordinating participant screening and randomization. Data analysis will be conducted by a study statistician blinded to participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT + MBRP (Experimental): Acceptance and Commitment Therapy + Mindfulness Based Relapse Prevention (ACT + MBRP) group will follow a manualized clinical protocol. Treatment will include 12 weekly group-based sessions, each lasting 90 minutes. Group sizes will range from 3 to 8. ACT + MBRP will be delivered via the VA Video Connect telehealth platform.
  Interventions: Behavioral: ACT+MBRP
- Education Control (EC) (Active Comparator): The EC group will follow a protocol that combines opioid education sessions and psychology-led pain education sessions that are offered as part of the interdisciplinary pain program. Specifically, education will include 12 group-based sessions, each lasting 60 to 90 minutes. Group sizes will range from 3 to 8. EC will be delivered via the VA Video Connect telehealth platform.
  Interventions: Behavioral: Education control

INTERVENTIONS:
Behavioral: ACT+MBRP — Intervention is behavioral treatment group that combines Acceptance and Commitment Therapy (ACT) with Mindfulness-Based Relapse Prevention. The group focuses on living with long-term pain, ways to complete daily living activities when you experience pain, coping with opioid and other drug cravings, and training in mindfulness practices.
  Arms: ACT + MBRP
Behavioral: Education control — Education control is behavioral treatment group that combines pain patient education with opioid and other drug education. The group focuses on experiences of long-term pain, instructions on how to function with this pain, and facts about opioids and other drugs.
  Arms: Education Control (EC)

SUMMARY:
This trial will recruit veterans with chronic pain (N = 160) who are prescribed buprenorphine for the treatment of opioid use disorder (OUD). We seek to: (1) examine the efficacy of an integrated treatment to reduce pain interference (Acceptance and Commitment Therapy and Mindfulness-Based Relapse Prevention [ACT + MBRP]) compared to an education control (EC) consisting of a protocol-based series of education sessions concerning chronic pain, opioids, and buprenorphine use and (2) examine how theoretically-relevant treatment mechanisms of pain acceptance, engagement in values-based action, and opioid craving are related to treatment outcomes. Interventions will be delivered via the VA Video Connect telehealth modality.

DETAILED DESCRIPTION:
There is compelling data that chronic pain and hazardous opioid use, considered individually, are significant and costly healthcare burdens in both veteran and nonveteran populations in the United States (US). When these two diagnoses are considered together, they appear to occur in a clinically significant proportion of patients. Further, opioid use disorder (OUD) interferes with chronic pain treatment outcomes and continued pain interferes with OUD outcomes treatment. While buprenorphine is effective for the treatment of pain and OUD, retention, relapse, and continued pain interference is not addressed through treatment with buprenorphine alone. Integrated treatments that target the key outcomes for both conditions, specifically pain's interference on functioning and opioid misuse/relapse, as developed in our prior work, allows for a parsimonious and efficacious way of providing treatment. Our recently completed pilot study indicated that such an integrated treatment was feasible and more effective than treatment as usual. To study this further, a multisite clinical trial comparing a three month integrated behavioral treatment that combines Acceptance and Commitment Therapy and Mindfulness-Based Relapse Prevention, as compared to an education control will be conducted with 160 veterans recruited from three VA Health Care Systems who have been stabilized on buprenorphine for the treatment of OUD. To assess longer-term outcomes, participants will be followed for 1 year after completion of the 3 month intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Stabilized on a dose of buprenorphine for a period of at least 1 month and less than six months. Buprenorphine stabilization will be defined as a consistent dose for at least 30 consecutive days.
2. Willing to comply with all study procedures and be available for the duration of the study
3. Male or female, aged 21 to 75 years.
4. Enrolled as a patient in one of the participating VA Co-Occurring Disorders clinics.
5. Presence of chronic pain for > 6 months in duration.

Exclusion Criteria:

1. Current or past diagnosis of schizophrenia, delusional disorder, psychotic or dissociative disorders.
2. Unable to read English.
3. Have a substance use disorder requiring a higher level of care than outpatient treatment (e.g., severe alcohol use disorder requiring inpatient detoxification).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain interference | Post-Treatment (month 3)
  Patient Reported Outcome Measurement Information System (PROMIS) Bank v1.0 Pain Interference- The National Institutes of Health (NIH) PROMIS toolkit measure for pain interference will be assessed via 8 items.

SECONDARY OUTCOMES:
Pain intensity | Post-Treatment (month 3)
  Pain intensity, including current and least/most/usual over the past week, will be assessed via a 0 (no pain) to 10 (maximum possible pain) Numerical Rating Scale.
Change in pain intensity | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Pain intensity, including current and least/most/usual over the past week, will be assessed via a 0 (no pain) to 10 (maximum possible pain) Numerical Rating Scale.
Opioid misuse | Post-Treatment (month 3)
  Current Opioid Misuse Measure (COMM) - The COMM measures opioid misuse risk and opioid-related behaviors via 17 items.
Depression | Post-Treatment (month 3)
  Patient Health Questionnaire 9 (PHQ-9) - The PHQ-9 will be used to assess depression via 9 self-report items.
Change in depression | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Patient Health Questionnaire 9 (PHQ-9) - The PHQ-9 will be used to assess depression via 9 self-report items.
Pain-related Fear | Post-Treatment (month 3)
  Pain Anxiety Symptom Scale (PASS) - Pain-related fear is reliably related to increased pain-related distress and disability via 20 self-report items.
Change in pain-related Fear | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Pain Anxiety Symptom Scale (PASS) - Pain-related fear is reliably related to increased pain-related distress and disability via 20 self-report items.
Alcohol and other drug use | Post-Treatment (month 3)
  Substance use over the past 7 days will be assessed via the Timeline Followback. Number of drinking days, number of days misusing substances, number of days of polysubstance use (using more than one substance), and drinks per drinking day will be calculated based on the number of days of drinking, number of days of substance misuse (where substance misuse is defined as non-prescribed opioids, non-prescribed other prescription drugs, illicit substances, and heavy drinking (4 or more drinks for women, 5 or more drinks for men)), and number of days of polysubstance use (defined as using more than one substance).
Change in alcohol and other drug use | Monthly.
  Substance use over the past 7 days will be assessed via the Timeline Followback. Number of drinking days, number of days misusing substances, number of days of polysubstance use (using more than one substance), and drinks per drinking day will be calculated based on the number of days of drinking, number of days of substance misuse (where substance misuse is defined as non-prescribed opioids, non-prescribed other prescription drugs, illicit substances, and heavy drinking (4 or more drinks for women, 5 or more drinks for men)), and number of days of polysubstance use (defined as using more than one substance).
Change in Pain interference | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Patient Reported Outcome Measurement Information System (PROMIS) Bank v1.0 Pain Interference- The National Institutes of Health (NIH) PROMIS toolkit measure for pain interference will be assessed via 8 items.
Change in opioid misuse | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Current Opioid Misuse Measure (COMM) - The COMM measures opioid misuse risk and opioid-related behaviors via 17 items.

OTHER OUTCOMES:
Social role functioning | Post-Treatment (month 3)
  PROMIS, Social Role Functioning via 8 self-report items.
Change in social role functioning | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  PROMIS, Social Role Functioning via 8 self-report items.
Psychosocial Impact of Illness | Post-Treatment (month 3)
  PROMIS, Psychosocial Impact of Illness via 8 self-report items
Change in psychosocial Impact of Illness | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  PROMIS, Psychosocial Impact of Illness via 8 self-report items
Physical Functioning | Post-Treatment (month 3)
  PROMIS, Physical Functioning via 6 self-report items
Change in Physical Functioning | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  PROMIS, Physical Functioning via 6 self-report items
Alcohol Use | Post-Treatment (month 3)
  Alcohol Use Disorders Identification Test, 10 self-report items
Change in Alcohol Use | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Alcohol Use Disorders Identification Test, 10 self-report items
Post-Traumatic Disorder Symptoms | Post-Treatment (month 3)
  PTSD Checklist-5, 20 self-report items
Change in Post-Traumatic Disorder Symptoms | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  PTSD Checklist-5, 20 self-report items
Generalized Anxiety | Post-Treatment (month 3)
  Generalized Anxiety Disorders Test (GAD-7), 7 self-report items
Change in Generalized Anxiety | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Generalized Anxiety Disorders Test (GAD-7), 7 self-report items
Sleep Disturbance | Post-Treatment (month 3)
  PROMIS, Sleep Disturbance via 6 items
Change in Sleep Disturbance | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  PROMIS, Sleep Disturbance via 6 items
Pain Catastrophizing | Post-Treatment (month 3)
  Pain Catastrophizing Scale - Short Form, 6 self-report items
Change in Pain Catastrophizing | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Pain Catastrophizing Scale - Short Form, 6 self-report items
Substance use | Post-Treatment (month 3)
  Tobacco, Alcohol, Prescription medication, and other Substance use Tool, 5 self-report items
Change in Substance use | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Tobacco, Alcohol, Prescription medication, and other Substance use Tool, 5 self-report items
Patient Global Impression of Change | Post-Treatment (month 3)
  Patient Global Impression of Change (PGIC) is a one item measure that reflects a patient's belief about the efficacy of treatment on a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Change in Patient Global Impression of Change | Pretreatment (month 0), post-treatment (month 3), and 6 and 12 month follow ups
  Patient Global Impression of Change (PGIC) is a one item measure that reflects a patient's belief about the efficacy of treatment on a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - San Francisco VA Health Care System, San Francisco, California
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Puget Sound VA Healthcare System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
It is expected that all data collected by award recipients and their collaborators, as part of the NIH Helping to End Addiction Long-term (HEAL) Initiative, will be shared with the NIH HEAL Initiative central data platform. Institutions who receive Data and/or Materials from this award for performance of activities under this award are required to use the Data and/or Materials only as outlined by the NIH HEAL Initiative, in a manner that is consistent with applicable state and federal laws and regulations, including any informed consent requirements and the terms of the institution's NIH funding.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the time of publication of the primary manuscript, or within 12 months of last patient procedure
Access Criteria: Implementation of the plan will follow the HEAL Public Access and Data Sharing Policy
URL: https://heal.nih.gov/about/public-access-data

REFERENCES:
- [Background] Vowles KE, Witkiewitz K, Cusack KJ, Gilliam WP, Cardon KE, Bowen S, Edwards KA, McEntee ML, Bailey RW. Integrated Behavioral Treatment for Veterans With Co-Morbid Chronic Pain and Hazardous Opioid Use: A Randomized Controlled Pilot Trial. J Pain. 2020 Jul-Aug;21(7-8):798-807. doi: 10.1016/j.jpain.2019.11.007. Epub 2019 Nov 21. PMID 31760109
- [Derived] Vowles KE, Witkiewitz K, Clarke E, Schmidt Z, Borsari B, Edwards KE, Korecki JR, Moniz-Lewis DI, Bondzie JA, Mullins C, Thoreson CI, Delacruz J, Wilkins CH, Nelson S, Delventura J, Henderson R, Katz A, Hua W, Watson E, Baxley C, Canlas BR, Pendleton T, Herbst E, Batki S. Rationale and design of a multisite randomized clinical trial examining an integrated behavioral treatment for veterans with co-occurring chronic pain and opioid use disorder: The pain and opioids integrated treatment in veterans (POSITIVE) trial. Contemp Clin Trials. 2023 Mar;126:107096. doi: 10.1016/j.cct.2023.107096. Epub 2023 Jan 21. PMID 36693589
- See also: Description of ACT+MBRP integrated treatment being tested in the current study. — https://doi.org/10.1016/j.jpain.2019.11.007